CLINICAL TRIAL: NCT00689468
Title: Echinacea Purpurea and Cranial Osteopathic Manipulative Treatment in Children With Recurrent Otitis Media: a Randomized Controlled Trial.
Brief Title: Echinacea Purpurea and Osteopathy in Children With Recurrent Otitis Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Richard Wahl, MD, Department of Pediatrics, University of Arizona
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Arizona HSC #98-83; NIH P50 HL61212-01
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-05

CONDITIONS: Otitis Media
Keywords: Otitis media; Echinacea; Osteopathic Medicine
MeSH Terms: conditions — Otitis Media | interventions — Echinacea extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): Osteopathic sham treatment plus placebo "Echinacea" drops
  Interventions: Procedure: Sham osteopathic manipulative treatment; Dietary Supplement: "Echinacea purpurea" placebo
- 2 (Active Comparator): Active Echinacea drops plus sham osteopathic treatment
  Interventions: Dietary Supplement: Echinacea purpurea; Procedure: Sham osteopathic manipulative treatment
- 3 (Active Comparator): Active osteopathic manipulation plus placebo "Echinacea" drops
  Interventions: Procedure: Cranial osteopathic manipulative treatment.; Dietary Supplement: "Echinacea purpurea" placebo
- 4 (Active Comparator): Active osteopathic manipulation plus active Echinacea drops.
  Interventions: Procedure: Cranial osteopathic manipulative treatment.; Dietary Supplement: Echinacea purpurea

INTERVENTIONS:
Procedure: Cranial osteopathic manipulative treatment. — A series of five cranial osteopathic manipulative treatment sessions scheduled over three months, and provided by osteopathic physicians whose practices are limited to osteopathic manipulative treatment. Treatment modalities were limited to cranial osteopathy, balanced membranous/ligamentous tension, and/or myofascial release (applied directly or indirectly).
  Arms: 3; 4
Dietary Supplement: Echinacea purpurea — 1:1 weight-to-volume 50% ethanol liquid extract of the fresh roots and dried mature seeds of Echinacea purpurea. Dosage: 0.5 ml orally 3 times daily for 3 days at the onset of cold symptoms, followed by 0.25 ml orally 3 times daily for 7 more days.
  Arms: 2; 4
Procedure: Sham osteopathic manipulative treatment — Sham osteopathic treatment consisted of a series of five osteopathic examinations only (palpation of the cranial bones and muscles and other structures) without treatment maneuvers.
  Arms: 1; 2
Dietary Supplement: "Echinacea purpurea" placebo — An identically labeled placebo contained 50% ethanol, 45% filtered water, food coloring and thickeners. Dosage: 0.5 ml orally 3 times daily for 3 days at the onset of cold symptoms, followed by 0.25 ml orally 3 times daily for 7 more days.
  Arms: 1; 3

SUMMARY:
This study was designed to evaluate the efficacy of the herb Echinacea purpurea and of cranial osteopathic manipulative treatment to prevent otitis media (middle ear infections) in young children.

DETAILED DESCRIPTION:
The use of complementary and alternative therapies by parents of young children remains common despite the lack of clinical trials demonstrating either the efficacy or safety of these treatments. Two of the more common complementary therapies used in young children with a history of recurrent otitis media are preparations of the herb Echinacea purpurea and cranial osteopathic manipulative treatment. This study represents one of the first double-blinded, placebo controlled trials of each approach in a population of young children who presented with three or more recent episodes of acute otitis media.

ELIGIBILITY:
Inclusion Criteria:

* 3 or more separate episodes of acute otitis media within a 6 month period, or
* 4 episodes of acute otitis media in one year,

Exclusion Criteria:

* Congenital malformations of the ears, nose, or throat
* Known or suspected allergy to echinacea
* Immune deficiency including HIV infection
* Tuberculosis
* Current use of prophylactic antibiotics
* Tympanostomy tubes in place
* Unwillingness of child to participate

Ages: 12 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 1999-07; Primary Completion 2002-09 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
The occurrence of a first episode of acute otitis media during the study period. | Six months

SECONDARY OUTCOMES:
The total number of episodes of diagnosed acute otitis media during the study period. | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Wahl, MD, Principal Investigator — University of Arizona; Michael B Aldous, MD, MPH, Principal Investigator — University of Arizona
Locations (3):
- United States (3):
  - Pediatric Osteopathic Center, Tucson, Arizona
  - KateCare Osteopathic Center, Tucson, Arizona
  - Pediatric Clinic, Arizona Health Sciences Center, Tucson, Arizona

REFERENCES:
- [Background] Mark JD, Grant KL, Barton LL. The use of dietary supplements in pediatrics: a study of echinacea. Clin Pediatr (Phila). 2001 May;40(5):265-9. doi: 10.1177/000992280104000505. PMID 11388676